CLINICAL TRIAL: NCT00788333
Title: A Phase I/II Trial of BMS-754807 in Combination With Trastuzumab (Herceptin®) in Subjects With Advanced or Metastatic Her-2-positive Breast Cancer
Brief Title: Combination Study of BMS-754807 and Herceptin® in Patients With Advanced or Metastatic Her-2-positive Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA191-004; EUDRACT #: 2009-013766-78
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: Advanced or Metastatic Her-2-positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — BMS 754807; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Combination
  Interventions: Drug: BMS-754807; Drug: trastuzumab (Herceptin®)

INTERVENTIONS:
Drug: BMS-754807 — Tablets, Oral, Dose escalation to MTD, then MTD to response/EOT, once daily, Varies - treatment is continued to disease progression or MD/subject/Sponsor decision to stop
  Other Names: IGF-IR
Drug: trastuzumab (Herceptin®) — IV solution, IV, 4mg/kg Day 1 loading dose, 2mg/kg once weekly, Varies - treatment is continued to disease progression or MD/subject/Sponsor decision to stop
  Other Names: Herceptin®

SUMMARY:
This is a Phase I/II study to evaluate the safety profile, tolerability, pharmacokinetics and pharmacodynamics following daily oral doses of 50 to 200 mg of BMS-754807 in combination with trastuzumab (Herceptin®) in subjects with advanced or metastatic Her-2-positive breast cancer. In addition, the study is expected to identify the recommended dose or dose range of BMS-754807 in combination with trastuzumab for Phase II studies and provide preliminary evidence of anti-tumor activity in Her-2-positive breast cancer subjects after trastuzumab failure

ELIGIBILITY:
For additional information on this trial, please call (910) 558-2913

Inclusion Criteria:

* Subjects with locally advanced or metastatic Her-2-positive breast cancer who have failed at least one trastuzumab containing regimen. Prior treatment with other Her-2-targeted agents (e.g. lapatinib, pertuzumab, trastuzumab DM-1 etc.) is allowed
* Histologic or cytologic diagnosis of Her-2-positive breast cancer
* ECOG status 0 - 1

Exclusion Criteria:

* Symptomatic brain metastasis
* Any condition requiring chronic use of steroids
* Any disorder with dysregulation of glucose homeostasis (history of Type 1 or 2 Diabetes Mellitus or prediabetic symptoms
* History of glucose intolerance
* Women of child-bearing potential unwilling or unable to use acceptable contraception methods

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
The dose escalation portion will determine the MTD and recommended Phase 2 dose or dose range of BMS-754807 when administered orally on a daily schedule in combination with trastuzumab administered at standard doses IV on a weekly basis | Every 30 days until MTD is reached

SECONDARY OUTCOMES:
Assess anti-tumor activity of combination at MTD of BMS-754807 (dose expansion cohort) | Every 8 weeks
Evaluate safety and tolerability of the combination regimen | Ongoing
Assess effect of combination therapy on glucose metabolism | At 30 days, then every 8 weeks
Explore whether co-medication with oral anti-hyperglycemic agent can enable adequate tolerability of the combination therapy if BMS-754807 induces hyperglycemia | Ongoing
Obtain BMS-754807 plasma concentrations vs time data for future population PK analysis | Days, 1,8,15,22

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (9):
- Australia (3):
  - Local Institution, Kurralta Park, South Australia
  - Local Institution, Frankston, Victoria
  - Local Institution, Geelong, Victoria
- Local Institution, Brussels, Belgium
- Canada (2):
  - Local Institution, Ottawa, Ontario
  - Local Institution, Toronto, Ontario
- Hungary (2):
  - Local Institution, Budapest
  - Local Institution, Miskolc
- Local Institution, Newcastle upon Tyne, Tyne and Wear, United Kingdom

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx